CLINICAL TRIAL: NCT04432402
Title: Efficacy and Safety of Lenalidomide in Combination With R-GemOx in First-line Treatment of Elderly Diffuse Large B Cell Lymphoma
Brief Title: Lenalidomide in Combination With R-GemOx in First-line Treatment of Elderly Diffuse Large B Cell Lymphoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, WEI XU, Professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-SR-443
Record Dates: First submitted 2020-06-11; First posted 2020-06-16 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: R-Gemox; Lenalidomide
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Lenalidomide; Rituximab; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lenalidomide in Combination With R-GemOx (Experimental): Lenalidomide 10mg、15mg、20mg、25mg qd PO d1-7 Rituximab 375mg/m2 ivd d0 Gemcitabine 1g/m2 ivd d1 Oxaliplatin 100mg/m2 ivd d1 every14 days as a cycle
  Interventions: Drug: Lenalidomide

INTERVENTIONS:
Drug: Lenalidomide — Lenalidomide: 10mg、15mg、20mg、25mg qd PO day 1-7, Rituximab: 375 mg/m2 IV day0, Gemcitabine :1g/m2 IV day 1, oxaliplatin 100mg/m2 IV day1 (every 14 days as a cycle)
  Other Names: Rituximab, Gemcitabine, oxaliplatin

SUMMARY:
The purpose of this study is to investigate efficacy and safety of Lenalidomide in combination with R-GemOx as first-line treatment of elderly patients with Diffuse large B cell lymphoma.

DETAILED DESCRIPTION:
Gemcitabine and Oxaliplatin(GemOx) shows effective activity in patients with relapsed diffuse large-cell lymphoma and other solid tumors. The purpose of this study is to investigate efficacy and safety of Lenalidomide in combination with R-GemOx as first-line treatment of elderly patients with Diffuse large B cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. The histopathologic diagnosis was DLBCL (except primary mediastinal large B cell lymphoma, primary central lymphoma, HIV related lymphoma).
2. Age older than 70 years or older than 60 years with Eastern Cooperative Oncology Group(ECOG) performance status(PS) ≥ 2;
3. Expected survival ≥ 12 weeks;
4. At least a measurable or evaluable disease at the time of enrolment (diameter ≥1.5cm);
5. Understand and voluntarily sign an informed consent form, able to adhere to the study visit schedule and other protocol requirements;
6. All patients must agree to take effective contraceptive measures during the trial measures

Exclusion Criteria:

1. Active hepatitis B or hepatitis C virus infection, as well as acquired, congenital immune deficiency diseases, including but not limited to HIV infected persons
2. Patients known to have varicella or herpes zoster virus infection
3. Previous exposure to any anti-tumor therapy
4. Poor hepatic and/or renal function, unless these abnormalities were related to the lymphoma
5. Poor bone-marrow reserve, defined as neutrophil count less than 1.5×109/L or platelet count less than 75×109/L, unless caused by bone marrow infiltration
6. History of deep vein thrombosis (DVT) or pulmonary embolism (PE) within past 12 months
7. New York Heart Association class III or IV cardiac failure; or Ejection fraction less than 50%;or history of following disease in past 6 months: acute coronary syndrome#acute heart failure#severe ventricular arrhythmia
8. Central nervous system (CNS) or meningeal involvement
9. Known sensitivity or allergy to investigational product
10. Major surgery within three weeks
11. Patients receiving organ transplantation
12. Patients with secondary tumour, excluding cured (5 years without relapse) in situ Non-melanoma skin cancer. superficial bladder cancer, in situ cervical cancer, Gastrointestinal intramucous carcinoma and breast cancer
13. Presence of Grade III nervous toxicity within past two weeks
14. Active and severe infectious diseases
15. Any potential drug abuse, medical, psychological or social conditions which may disturb this investigation and assessment
16. In any conditions which investigator considered ineligible for this study.
17. Histologic transformation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2020-06-14 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose | at the end of the first cycle of R2-GemOx (each cycle is 14 days)
  Maximum tolerated dose
Dose limiting toxicity | 28 days
  Dose limiting toxicity
Dose limiting toxicity | 2 years
  Dose limiting toxicity

SECONDARY OUTCOMES:
progression-free survival | 2 years
  progression-free survival
overall survival | 2 years
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Wei Xu, M.D., Ph.D, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- The first Affiliated Hospital Of Nanjing Medical University(JiangSu Province Hospital), Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes